CLINICAL TRIAL: NCT05354791
Title: Comparison of Success and Injury (Neuropraxia) Rate When Performing the Sciatic Nerve Block in the Popliteal Fossa Pre vs. Post Spinal Anesthesia for Foot and Anke Procedures: Retrospective Review
Brief Title: Pre-post Spinal Popliteal Block
Status: Terminated | Type: Observational
Why Stopped: Retrospective study that the PI decided not to proceed with
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1642
Record Dates: First submitted 2022-04-08; First posted 2022-04-29 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Foot Surgery; Ankle Surgery
Keywords: lower extremity peripheral nerve block; spinal anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective chart review to determine the non-inferiority of performing lower extremity peripheral nerve block placement under spinal anesthesia compared to its pre-spinal counterpart.

DETAILED DESCRIPTION:
This is a retrospective chart review to determine the non-inferiority of performing lower extremity peripheral nerve block placement under spinal anesthesia compared to its pre-spinal counterpart.

Primary outcome:

- The investiigators will be looking into persistent abnormal neuropathic symptoms lasting more than 7 days following a sciatic popliteal nerve block.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory foot surgery
* ambulatory ankle surgery
* use of spinal Anesthesia
* use of pre-spinal anesthesia nerve block techniques
* use of sciatic nerve block

Exclusion Criteria:

* all other surgeries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to analyze data for patients who underwent ambulatory foot or ankle procedures with the use of spinal anesthesia and sciatic nerve block in the popliteal fossa at HSS between March 1, 2016 and February 24, 2020
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Persistent Abnormal Neuropathic Symptoms | lasting more than 7 days following a sciatic popliteal nerve block
  Definition of abnormal neuropathic symptoms including numbness, tingling, burning, or pain sensation.

SECONDARY OUTCOMES:
NRS pain scores in recovery | PACU recovery stay (up to 48 hours)
  A score on a scale from 0 to 10 on how bad the pain is. 0 means no pain, 10 means worst pain. A lower score means a better outcome.
Amount of supplemental analgesic and antiemetic provided in the PACU | PACU recovery stay (up to 48 hours)
  This includes: IV dilaudid push, oral oxycodone, tramadol, hydrocodone, dilaudid, acetaminophen, ketorolac, ondansetron, dexamethasone.
Anesthesia induction time | From the time which patients enter the OR to time of anesthesia induction end (up to 24 hours)
  time from entering the OR to time of anesthesia induction end as defined by the completion of both the spinal and sciatic nerve blockade
Number of hypoxemia events during induction time | during induction time (up to 24 hours)
Amount of sedation given | during induction time (up to 24 hours)
  fentanyl, ketamine, midazolam, propofol

CONTACTS AND LOCATIONS:
Overall Officials: Sang Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States